CLINICAL TRIAL: NCT03769259
Title: Brief Cognitive Behavioral Therapy Replication Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Ohio State University (Other); Lowcountry Center for Veterans Research (Unknown); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Craig Bryan, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMCCL.2018.0009; W81XWH1820022 (Other Grant/Funding Number: U.S. Army Medical Research Acquisition Activity)
Record Dates: First submitted 2018-11-01; First posted 2018-12-07 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Suicide, Attempted; Suicidal Ideation
Keywords: suicide; suicidal ideation; ambivalence; suicide ambivalence; reasons for living; reasons for dying; military; clinical trial; cognitive behavioral therapy; psychotherapy; crisis; Crisis Response Plan (CRP); Present Centered Therapy (PCT); Brief Cognitive-Behavioral Therapy (BCBT)
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation; Suicide | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Brief Cognitive Behavioral Therapy (BCBT); Behavioral: Treatment as Usual (TAU)
- Present-Centered Therapy (Active Comparator)
  Interventions: Behavioral: Present-Centered Therapy (PCT); Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Therapy (BCBT) — Participants in BCBT receive 12 outpatient individual psychotherapy sessions scheduled on a weekly or biweekly basis, with the first session lasting 90 minutes and subsequent sessions lasting 60 minutes. BCBT was is delivered in three sequential phases. In phase I (5 sessions), the therapist identifies patient-specific factors that contribute to and maintain suicidal behaviors, provides a cognitive-behavioral conceptualization, collaboratively develops a crisis response plan, and teaches basic emotion regulation skills. In phase II (5 sessions), the therapist applies cognitive strategies to reduce beliefs and assumptions that serve as vulnerabilities to suicidal behavior. In phase III (2 sessions), a relapse prevention task is conducted.
  Other Names: Cognitive Therapy
  Arms: Brief Cognitive Behavioral Therapy
Behavioral: Present-Centered Therapy (PCT) — Participants in PCT will receive will include 12 outpatient individual psychotherapy sessions scheduled on a weekly or biweekly basis, with the first session lasting 90 minutes and subsequent sessions lasting 60 minutes. PCT consists of (1) psychoeducation about the typical symptoms and features associated with suicidal thoughts and behaviors among military personnel; (2) normalization of symptoms; (3) experience of receipt of support and feedback from a licensed professional; and (4) positive interpersonal interactions.
  Arms: Present-Centered Therapy
Behavioral: Treatment as Usual (TAU) — All participants will receive the following interventions or procedures, regardless of treatment assignment:
  * Suicide risk assessment using the Columbia Suicide Severity Rating Scale
  * VA's safety planning intervention, which include Military Crisis Line contact information and lethal means access reduction
  * Caring contacts and outreach
  * Psychotropic medication, group therapy, substance abuse counseling, and other mental health interventions provided routinely as a part of treatment as usual

SUMMARY:
The overall goal for the proposed project is to test the effectiveness of BCBT for the prevention of suicide attempts in a sample of treatment-seeking U.S. military personnel and veterans. The standard null hypothesis will involve tests conducted comparing improvement following BCBT (treatment duration of 12 weeks) to Person-Centered Therapy (PCT). The primary outcome comparisons will include direct markers of suicidality (i.e. suicide, suicide attempts). Secondary outcomes will be suicide ideation and indicators of psychiatric distress (e.g., depression, hopelessness). We also aim to assess several hypothesized psychological and neurocognitive mediators of treatment effects (e.g., wish to live, attentional bias, emotion regulation). Participants will be followed for 2 years posttreatment by independent evaluators blind to treatment condition.

DETAILED DESCRIPTION:
The number of suicides by military personnel and veterans has steadily increased during the past few decades and remains elevated. Previous research conducted with active duty Army personnel supports the superiority of BCBT and its components over treatment as usual for the reduction of suicide attempts. Additional research is needed to determine if these effects are generalizable to military personnel and veterans more broadly and to confirm hypothesized mechanisms of action. Reference to "active duty" refers to U.S. military service members that have been activated and deployed as a part of Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF) in accordance with federal orders under Title 10 or 32, United States Code. Reference to "veteran" refers to any person who has served in the U.S. military at any time, regardless of Branch, Component, era, or discharge status.

Specific Aim 1:To replicate previous findings supporting the efficacy of BCBT for the prevention of suicide attempts among military personnel and veterans (regardless of Axis I or II diagnosis). The standard null hypothesis will involve tests conducted comparing improvement following BCBT to Present-Centered Therapy (PCT)

Specific Aim 2: To identify cognitive-affective mediators of BCBT's effects on risk for suicide attempt.

ELIGIBILITY:
Inclusion Criteria:

* Current or past service in the U.S. military
* 18 years of age or older
* Reporting current suicide ideation with intent to die and/or a suicide attempt within the past two weeks
* Ability to understand and speak the English language; and ability to complete the informed consent process.

Exclusion Criteria:

* Psychiatric or medical condition that precludes the ability to provide informed consent or participation in outpatient treatment (e.g., psychosis, mania, acute intoxication).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in number of suicide attempts from baseline | Assessed every 3 months through study completion (average of 2 years)
  The change in number of suicide attempts from baseline will be assessed through review of participants' medical records and through participants' responses to the Self-Injurious Thoughts and Behaviors Interview. The Self-Injurious Thoughts and Behaviors Interview is a structured interview assessing history of suicidal thoughts and behaviors, including suicide attempt history (dates, methods, and severity (e.g., need for medical attention) of previous suicide attempts). An increased number of suicide attempts at any assessment is considered a worse outcome.

SECONDARY OUTCOMES:
Change in suicidal ideation scores from baseline | Assessed once per week until completion of treatment (average of 12 weeks) and at every 3 months through study completion (average of 2 years)
  The Beck Scale for Suicide Ideation is a 21-item self-report measure of the severity of current suicidal ideation. Items 1-19 measure current suicidal ideation, with summed total scores for these items ranging from 0-38. Higher scores are associated with more severe suicidal ideation and are considered a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Craig J Bryan, PsyD, ABPP, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Naval Medical Center Camp Lejeune, Jacksonville, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Lowcountry Center for Veterans Research, Charleston, South Carolina

REFERENCES:
- [Background] Bryan CJ, Rudd MD, Wertenberger E. Reasons for suicide attempts in a clinical sample of active duty soldiers. J Affect Disord. 2013 Jan 10;144(1-2):148-52. doi: 10.1016/j.jad.2012.06.030. Epub 2012 Aug 1. PMID 22858207
- [Background] Bryan CJ, Rudd MD. Life stressors, emotional distress, and trauma-related thoughts occurring in the 24 h preceding active duty U.S. soldiers' suicide attempts. J Psychiatr Res. 2012 Jul;46(7):843-8. doi: 10.1016/j.jpsychires.2012.03.012. Epub 2012 Apr 1. PMID 22464944
- [Background] Rudd MD, Bryan CJ, Wertenberger EG, Peterson AL, Young-McCaughan S, Mintz J, Williams SR, Arne KA, Breitbach J, Delano K, Wilkinson E, Bruce TO. Brief cognitive-behavioral therapy effects on post-treatment suicide attempts in a military sample: results of a randomized clinical trial with 2-year follow-up. Am J Psychiatry. 2015 May;172(5):441-9. doi: 10.1176/appi.ajp.2014.14070843. Epub 2015 Feb 13. PMID 25677353
- [Background] Bryan CJ, Mintz J, Clemans TA, Leeson B, Burch TS, Williams SR, Maney E, Rudd MD. Effect of crisis response planning vs. contracts for safety on suicide risk in U.S. Army Soldiers: A randomized clinical trial. J Affect Disord. 2017 Apr 1;212:64-72. doi: 10.1016/j.jad.2017.01.028. Epub 2017 Jan 23. PMID 28142085
- [Derived] Bryan CJ, Khazem LR, Baker JC, Brown LA, Taylor DJ, Pruiksma KE, Acierno R, Larick JG, Baucom BRW, Garland EL, Rudd MD. Brief Cognitive Behavioral Therapy for Suicidal Military Personnel and Veterans: The Military Suicide Prevention Intervention Research (MSPIRE) Randomized Clinical Trial. JAMA Psychiatry. 2025 Dec 1;82(12):1169-1176. doi: 10.1001/jamapsychiatry.2025.2850. PMID 41060644
- See also: Suicide and Trauma Reduction Initiative (STRIVE) — http://strive2be.org

DOCUMENTS (1):
  • Informed Consent Form (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT03769259/ICF_000.pdf